CLINICAL TRIAL: NCT06098911
Title: Comparative Clinical and Radiographic Evaluation of Casein Phosphopeptide Amorphous Calcium Phosphate Under Glass Ionomer in Atraumatic Restorative Treatment Versus Conventional Atraumatic Restorative Treatment in Primary Teeth: A Randomized Clinical Trial
Brief Title: Modified Atraumatic Restorative Treatment Using CPP ACP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Sherif, Dr. Mai Sherif, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPP ACP in ART
Record Dates: First submitted 2023-10-12; First posted 2023-10-25 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Caries
Keywords: CPP ACP; atraumatic restorative treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MI varnish (CPP ACP) under glass ionomer in ART group (Experimental): Application of a thin layer of casein phosphopeptide amorphous calcium phosphate ( CPP ACP ) varnish as indirect pulp capping material under glass-ionomer (Riva Light cure GC company ) in Atraumatic restorative technique.
  Interventions: Device: MI varnish
- Conventional ART (No Intervention): Placement of glass-ionomer restoration ( Riva Light Cure ) only in Atraumatic restorative technique.

INTERVENTIONS:
Device: MI varnish — delivers a powerful dose of fluoride, with the added booster effect of the calcium and phosphate ions through its patented Recaldent™ technology. High initial fluoride release. Minimizes tooth sensitivity and strengthens enamel. Neutral pH of 6,6 enhances enamel and dentin acid resistance and inhibits demineralization
  Other Names: CPP ACP
  Arms: MI varnish (CPP ACP) under glass ionomer in ART group

SUMMARY:
To evaluate the clinical and radiographic success of using Casein Phosphopeptide Amorphous Calcium Phosphate (CPP-ACP) under glass ionomer restorations in atraumatic restorative treatment as a biomimetic approach in pediatric dentistry.

DETAILED DESCRIPTION:
With the growing popularity of ART in the field of pediatric dentistry, a great deal of research has been done in recent years. Researchers are keen to explore the rich possibilities and variations of ART technique that can help doctors practice better and do more for their patients. Alternatives include detours to regenerative dentistry, which is becoming more and more popular these days.

CPP ACP is still of great interest in the region due to its remineralizing action. However, to our knowledge, clinical and radiological success involving tissue regeneration by CPP-ACP is understudied. Furthermore, the studies conducted justify the need for further research on the use of CPP-ACP as an indirect material under glass ionomers in ART. Therefore, this study aims to conclude whether CPP ACP has added value in regenerating, reducing pain, and improving repair retention in caries-affected dentin lesions.

ELIGIBILITY:
* Inclusion Criteria:

Clinical Criteria:

Children aged 4-7 years. Apparently healthy children. Children with mild to moderate occlusal carious lesions in the mandibular second primary molar indicated for indirect pulp capping.

No history of spontaneous pain, pathologic mobility, draining sinus tract, redness or swelling of vestibule.

Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.

Radiographic criteria:

* No sign of radiolucency in periapical or furcation area.
* No widening of PDL space or loss of lamina dura continuity.
* No evidence of internal/external pathologic root resorption.

Exclusion Criteria:

* Uncooperative children to avoid time waste and attrition bias.
* Children with systemic disease as some systemic diseases may have effect on the outcome Children with known allergy to any of the components being utilized. Molars near exfoliation.

Primary molars with more than half of the root resorbed or with periapical pathology as evident radiographically Mobile or ankylosed molars with no permanent successors

* Unable to attend follow-up visits to avoid attrition bias by decreasing number of drop off cases.
* Refusal of participation as the parent of child has the authority of participation.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 12 months
  Verbal question to the patient form score 0-5 where o is no pain and maximum pain indicates 5
Marginal integrity | 12 months
  Visual and clinical examination (by probe and mirror or any change in color or breakage of restoration, recurrent caries as direct observation) from score 0-5 where 0 gap free marginal interface, 1 indicates mircoleakage occur in 1 surface, 2 in 2 surfaces, 3 in 3 surfaces, 4 in 4 surfaces, 5 loss of whole restoration.

SECONDARY OUTCOMES:
Absence of furcation or periapical radiolucency | 12 months
  Intra oral periapical Xray
Absence of any internal or external root resorption | 12 months
  Intra oral periapical Xray

IPD SHARING:
Plan to Share IPD: No
Access to final data will be allowed to the operator (principal investigator) and the main and co-supervisors of the study, who aren't involved in assessing the outcome. All data sets will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded to any identifying participant information.

REFERENCES:
- [Result] Bresciani E. Clinical trials with Atraumatic Restorative Treatment (ART) in deciduos and permanent teeth. J Appl Oral Sci. 2006;14 Suppl:14-9. doi: 10.1590/s1678-77572006000700004. PMID 19089081
- See also: Alexandria university — https://adjalexu.journals.ekb.eg/article_271935_184e1fe67a975f7872c8e3b1b3e70e6b.pdf